CLINICAL TRIAL: NCT04474678
Title: A Quality Improvement Project to Implement Psychosocial Care Standards in Clinical Practice in Pediatric Oncology "My Logbook! - I Know my Way Around!" ("Mein Logbuch - Ich Kenne Mich Aus!") Development and Evaluation of a Consensus and Evidence Based Psychosocial Therapy Tool in a Preliminary Psychosocial Study on Therapy Optimization.
Brief Title: Quality Improvement Project - "My Logbook! - I Know my Way Around!"; ("Mein Logbuch - Ich Kenne Mich Aus!")
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Collaborators: St. Anna Kinderspital, Austria (Other); Charite University, Berlin, Germany (Other); Cnopfsche Kinderklinik, Nürnberg (Unknown); Kepler University Hospital (Other); University Hospital, Saarland (Other); Hannover Medical School (Other); Krankenhaus Bozen (Other); Goethe University (Other); Universitätsklinikum Hamburg-Eppendorf (Other); Universitätsklinikum Leipzig (Other); University Hospital Muenster (Other); University Hospital Tuebingen (Other); Salzburger Landeskliniken (Other); Leuwaldhof St.Veit (Kinder- und Jugendreha) (Unknown); University Hospital, Essen (Other); Medical University of Graz (Other); University Hospital Erlangen (Other); Wuerzburg University Hospital (Other); Klinik Bad Oexen, Germany (Unknown); Universitätsklinikum Köln (Other); University Hospital Schleswig-Holstein (Other); University Hospital Carl Gustav Carus (Other); Universitätsmedizin Mannheim (Other); University Hospital Regensburg (Other); Luca-Dethlefsen-Hilfe e.V. (Unknown); Insel Gruppe AG, University Hospital Bern (Other); Staedtisches Klinikum Karlsruhe (Other)
Responsible Party: Principal Investigator, Dr. Liesa J. Weiler-Wichtl, Project Coordinator, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1564/2017
Record Dates: First submitted 2020-06-23; First posted 2020-07-17 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Brain Tumor; Neurofibromatoses; Sarcoma; Leukemia; Hematologic Diseases; Neuroblastoma
MeSH Terms: conditions — Brain Neoplasms; Neurofibromatoses; Sarcoma; Leukemia; Hematologic Diseases; Neuroblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All Patients (Other): Since this is a single-group study, all patients are within the same arm
  Interventions: Other: "My Logbook! - I know my way around!"

INTERVENTIONS:
Other: "My Logbook! - I know my way around!" — Special issues/booklets of "My Logbook - I know my way around!" - Every booklet is based on evidence-based interventions. It illustrates psychosocial and interdisciplinary processes in a standardized way, resulting in a practical guide ("My Logbook") to accompany the child throughout all stages of oncological treatment.

SUMMARY:
In this study, the main goal is to implement and evaluate a novel, evidence-based psycho-educative program for children in oncological care. Patients are provided with booklets tailored to each specific stage of their treatment. Among other factors, children's emotional well-being is evaluated as well as feasibility. The study is carried out at multiple sites across Austria, Germany and Italy/South Tirol.

DETAILED DESCRIPTION:
It is well documented that the prevalence of mental disorders in childhood cancer survivors is twice to quadruple compared to healthy controls. Effects range from impaired emotional balance, fear of recidivisms, helplessness, depression to post traumatic stress disorder.

As a basis for interventions to preventively address these issues and moreover, to achieve defined psychosocial goals in the field of paediatric oncology, guidelines and standards systematically describe stressors and resources in particularly challenging situations. Nevertheless, despite these guidelines, actual care is quite heterogenous due to differences in setting, provision and profession. Studies show that integrated models of psychosocial care yield better outcomes. Integrated care systems can enhance patient satisfaction, increase perceived quality of care, and enable access to services and reduce service costs. Highly complex, system-wide interventions such as models of integrated care represent considerable challenges for operationalisation of relevant factors and evaluation of whole processes compared to single interventions (e.g. relaxation techniques). Quality improvement (QI) is an iterative process designed to make controlled changes within the health care delivery system to provide patients with high-quality care that meets both their expectations and needs. In terms of quality assurance, this QI Project aims to operationalize recommendations of the S3 guideline for psychosocial care which results in a combined process- and patient-oriented intervention and evaluation tool - bridging the gap between standards/evidence and clinical practice.

The "Onco-Mini-Version" of "My Logbook - I know my way around" already comprises a Starter-Kit and 8 booklets, which cover at least one main issue of every treatment phase: initial contact, medical assessment (MRI), supportive therapy (chemotherapy, radio therapy), rehabilitation and after-care. All interventions are carried out by a clinical psychologist or psychosocial staff specialized in pediatric psychooncology and are understood as part of an integrated care system. Every booklet provides practical materials with enhanced stimulating elements to encourage the child to explore actively. The booklets are structured in two face-to-face sessions covering psychoeducational, activity & practice and reflective aspects.

The core of this QI project is a multilevel and interdisciplinary approach characterized by iterative processes. PDSA (Plan, Do, Study, Act) cycles were applied in all steps of conceptualization and implementation of this project. It aims to systematically improve psychosocial care of pediatric cancer patients through being implemented in a large number of hospitals in the German-speaking world. The proposed multicenter pilot phase promotes emotional well-being and level of information of the child during treatment through transfer of knowledge and coping skills. Moreover, it addresses feasibility of the tool but also the impact of medical procedures on feasibility. In the long term, the program is intended to help attenuate psychological late effects of oncological conditions and their treatments.

ELIGIBILITY:
Inclusion Criteria experimental group:

* currently or formerly treated for oncological condition
* children/families at standard risk (Pediatric Psychosocial Preventative Health Model (PPPHM))
* at least average cognitive abilities (as measured via intelligence test)

Inclusion Criteria control group:

* currently or formerly treated for oncological condition

Exclusion Criteria:

* non-German speaking
* Major vision impairments
* Major auditive impairments

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 240 (Actual)
Dates: Start 2020-09-07 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Emotional well-being, T1 | Based on the medical therapy protocol, after medical consultation, prior to first session of the special issue (booklet) - through study completion or end of medical treatment, an average of 1 year
  Patients' emotional well-being is evaluated using a visual array of emotional displays. Patients can choose three emotions that describe their current situation best. For analysis, emotions are categorized into positive, neutral, and negative emotions. Emotional well-being is evaluated longitudinally over multiple points of time. The diagnostic tool was developed in-house, publication is pending.
Emotional well-being, T2 | Post to first session of the special issue (booklet) - through study completion or end of medical treatment, an average of 1 year
  Patients' emotional well-being is evaluated using a visual array of emotional displays. Patients can choose three emotions that describe their current situation best. For analysis, emotions are categorized into positive, neutral, and negative emotions. Emotional well-being is evaluated longitudinally over multiple points of time. The diagnostic tool was developed in-house, publication is pending.
Emotional well-being, T3 | During, but before completion of treatment; prior to second session of the special issue (booklet) - through study completion or end of medical treatment, an average of 1 year
  Patients' emotional well-being is evaluated using a visual array of emotional displays. Patients can choose three emotions that describe their current situation best. For analysis, emotions are categorized into positive, neutral, and negative emotions. Emotional well-being is evaluated longitudinally over multiple points of time. The diagnostic tool was developed in-house, publication is pending.
Emotional well-being, T4 | During, post to second session of the special issue (booklet) - through study completion or end of medical treatment, an average of 1 year
  Patients' emotional well-being is evaluated using a visual array of emotional displays. Patients can choose three emotions that describe their current situation best. For analysis, emotions are categorized into positive, neutral, and negative emotions. Emotional well-being is evaluated longitudinally over multiple points of time. The diagnostic tool was developed in-house, publication is pending.
Emotional well-being, T5 | During, but before completion of treatment - through study completion or end of medical treatment, an average of 1 year
  Patients' emotional well-being is evaluated using a visual array of emotional displays. Patients can choose three emotions that describe their current situation best. For analysis, emotions are categorized into positive, neutral, and negative emotions. Emotional well-being is evaluated longitudinally over multiple points of time. The diagnostic tool was developed in-house, publication is pending.
Knowledgeability, T1 | Based on the medical therapy protocol, after medical consultation, prior to first session of the special issue (booklet) - through study completion or end of medical treatment, an average of 1 year
  Patients are asked to rate their own knowledgeability regarding treatment, illness and hospital environment on a five-point scale ranging from "beginner" to "expert". Knowledgeability is evaluated longitudinally over multiple points of time. The diagnostic tool was developed in-house.
Knowledgeability, T2 | Post to first session of the special issue (booklet) - through study completion or end of medical treatment, an average of 1 year
  Patients are asked to rate their own knowledgeability regarding treatment, illness and hospital environment on a five-point scale ranging from "beginner" to "expert". Knowledgeability is evaluated longitudinally over multiple points of time. The diagnostic tool was developed in-house.
Knowledgeability, T3 | During, but before completion of treatment; prior to second session of the special issue (booklet) - through study completion or end of medical treatment, an average of 1 year
  Patients are asked to rate their own knowledgeability regarding treatment, illness and hospital environment on a five-point scale ranging from "beginner" to "expert". Knowledgeability is evaluated longitudinally over multiple points of time. The diagnostic tool was developed in-house.
Knowledgeability, T4 | During, post to second session of the special issue (booklet) - through study completion or end of medical treatment, an average of 1 year
  Patients are asked to rate their own knowledgeability regarding treatment, illness and hospital environment on a five-point scale ranging from "beginner" to "expert". Knowledgeability is evaluated longitudinally over multiple points of time. The diagnostic tool was developed in-house.
Knowledgeability, T5 | During, but before completion of treatment - through study completion or end of medical treatment, an average of 1 year
  Patients are asked to rate their own knowledgeability regarding treatment, illness and hospital environment on a five-point scale ranging from "beginner" to "expert". Knowledgeability is evaluated longitudinally over multiple points of time. The diagnostic tool was developed in-house.
Feasibility of program | Feasibility of program is evaluated following the second session which on average takes place one to six months after start of the treatment of the special issue (booklet). - through study completion or end of medical treatment, an average of 1 year
  Rating of feasibility of the program by medical staff

SECONDARY OUTCOMES:
Intelligence test | During the first two months from diagnosis or start of psychosocial treatment - up to three Months
  Patients are administered a standardized intelligence test, dependent on their age, e.g.
  Wechsler Intelligence Scale for Children IV WISC-IV, Petermann & Petermann, 2014 or other comparable methods due to clinical standards
Strengths and Difficulties Questionnaire (SDQ; Goodman, 1999) | During the first two months from diagnosis or start of psychosocial treatment - up to three Months
  The Strengths and Difficulties Questionnaire (SDQ) is a brief behavioural screening questionnaire about 3-16 year olds.
KINDLR (Ravens-Sieberer & Bullinger, 2000) | During the first two months from diagnosis or start of psychosocial treatment - up to three Months
  The KINDLR is a standardized questionnaire for the assessment of quality of life in children and adolescents.
Questionnaire on Health Competence in Children and Adolescents, (Weiler, Fohn, Pletschko, Schwarzinger, & Leiss, 2017) | During the first two months from diagnosis or start of psychosocial treatment - up to three Months
  Questionnaire for the assessment of health competence in children and adolescents
Medical information | Within the first week of treatment - up to three Months
  Diagnosis, date of diagnosis, pre-existing conditions, secondary conditions, form of treatment/therapy, psychiatric diagnoses, neurological status
Demographic data | During the first two months from diagnosis or start of psychosocial treatment - up to three Months
  Age of patient, sex, parents' education, parents' profession, school form, mother language of patient

CONTACTS AND LOCATIONS:
Locations (22):
- Austria (5):
  - Rehabilitationszentrum St. Veit im Pongau, Sankt Veit im Pongau, Salzburg
  - Kepler Universitätsklinikum, Linz, Upper Austria
  - Medical University Graz, Graz
  - Medical University of Vienna, Vienna
  - St. Anna Kinderspital, Vienna
- Germany (15):
  - Universitätsklinikum Frankfurt am Main, Frankfurt am Main, Hesse
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - Universitätsklinikum Essen, Essen, North Rhine-Westphalia
  - Universitätsklinikum Münster, Münster, North Rhine-Westphalia
  - Universitätsklinikum des Saarlandes, Homburg, Saarland
  - Universitätsklinikum Leipzig, Leipzig, Saxony
  - Klinik Bad Oexen, Bad Oeynhausen
  - Charité - Universitätsmedizin Berlin, Berlin
  - Luca-Dethlefsen-Hilfe e.V., Bielefeld
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Universitätsklinikum Mannheim, Mannheim
  - Universitätsklinikum Regensburg, Regensburg
  - Universitätsklinikum Tübingen, Tübingen
  - Universitätsklinikum Würzburg, Würzburg
- Ospedale di Bolzano, Bolzano, Trentino-Alto Adige, Italy
- Inselspital, Universitätsspital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kazak AE, Abrams AN, Banks J, Christofferson J, DiDonato S, Grootenhuis MA, Kabour M, Madan-Swain A, Patel SK, Zadeh S, Kupst MJ. Psychosocial Assessment as a Standard of Care in Pediatric Cancer. Pediatr Blood Cancer. 2015 Dec;62 Suppl 5:S426-59. doi: 10.1002/pbc.25730. PMID 26700916
- [Background] Scialla MA, Canter KS, Chen FF, Kolb EA, Sandler E, Wiener L, Kazak AE. Delivery of care consistent with the psychosocial standards in pediatric cancer: Current practices in the United States. Pediatr Blood Cancer. 2018 Mar;65(3):10.1002/pbc.26869. doi: 10.1002/pbc.26869. Epub 2017 Oct 28. PMID 29080381
- [Background] Baxter S, Johnson M, Chambers D, Sutton A, Goyder E, Booth A. The effects of integrated care: a systematic review of UK and international evidence. BMC Health Serv Res. 2018 May 10;18(1):350. doi: 10.1186/s12913-018-3161-3. PMID 29747651
- [Background] Schurman JV, Gayes LA, Slosky L, Hunter ME, Pino FA. Publishing quality improvement work in Clinical Practice in Pediatric Psychology: The "why" and "how to". Clinical Practice in Pediatric Psychology. 2015 Mar; 3(1):80.
- [Background] Schröder HM, Lilienthal S, Schreiber-Gollwitzer BM, Griessmeier B, Leiss U. Psychosoziale Versorgung in der Pädiatrischen Onkologie und Hämatologie. PSAPOH (Hg.). 2013.
- [Background] Stuber ML, Meeske KA, Krull KR, Leisenring W, Stratton K, Kazak AE, Huber M, Zebrack B, Uijtdehaage SH, Mertens AC, Robison LL, Zeltzer LK. Prevalence and predictors of posttraumatic stress disorder in adult survivors of childhood cancer. Pediatrics. 2010 May;125(5):e1124-34. doi: 10.1542/peds.2009-2308. PMID 20435702
- [Background] Koch U, Mehnert A, Harter M. [Chronic somatic disorders and psychological comorbidity]. Bundesgesundheitsblatt Gesundheitsforschung Gesundheitsschutz. 2011 Jan;54(1):1-3. doi: 10.1007/s00103-010-1196-7. No abstract available. German. PMID 21246321
- [Derived] Weiler-Wichtl LJ, Fohn-Erhold V, Rosenmayr V, Hansl R, Hopfgartner M, Pal-Handl K, Wasinger-Brandweiner V, Herzog K, Neumann K, Schellenberg T, Schonenberger-Loppacher D, Faist-Schweika C, Schonthaler B, Budich M, Stember N, Wiegele K, Reddig M, Paduch A, Lein-Kohler I, Gorgen S, Wienands H, Gauf H, Hoffmann R, Kollmann A, Just U, Salzmann N, Neunsinger P, Gerhardt M, Essl S, Borbely J, Kopper M, Rinner S, Schubert L, Leiss U. Benefits of applying standardized frameworks to implement psychosocial tools such as the 'My Logbook'. Support Care Cancer. 2024 Nov 14;32(12):789. doi: 10.1007/s00520-024-08981-7. PMID 39538073
- [Derived] Weiler-Wichtl LJ, Fohn-Erhold V, Rosenmayr V, Hansl R, Hopfgartner M, Fries J, Schneider C, Herzog K, Schellenberg T, Schonthaler B, Stember N, Lein-Kohler I, Hoffmann R, Kollmann A, Salzmann N, Essl S, Pal-Handl K, Wasinger-Brandweiner V, Rinner S, Schubert L, Lange S, Leiss U. Preparing Children for Invasive Medical Cancer Treatment with "My Logbook": Preliminary Results of a Pilot Study. J Cancer Educ. 2025 Feb;40(1):132-141. doi: 10.1007/s13187-024-02481-2. Epub 2024 Aug 7. PMID 39107671